CLINICAL TRIAL: NCT07268352
Title: The Effect of Ventilation Frequency on Diaper Dermatitis Recovery and Maternal Self-Efficacy in Infants Aged 0-3 Months: A Randomized Controlled Trial
Acronym: Diaper Dermati
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Shahla Shafaati Laleh, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SSL&AYK
Record Dates: First submitted 2025-11-16; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Family-centered Care
Keywords: Diaper dermatitis; ventilation; maternal self-efficacy; infant care; randomized controlled trial.
MeSH Terms: conditions — Diaper Rash; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: "Diaper-Free Ventilation: 5 Minutes, 6 Times Daily (Active Comparator): This arm of the study focuses on providing infants with diaper-free air exposure as a method to improve recovery from diaper dermatitis. In this group, participants are given the opportunity to be without a diaper for a duration of 5 minutes, and this process is repeated six times throughout the day.
  Interventions: Behavioral: Diaper-Free Air Exposure Protocol"
- Group B: "Diaper-Free Ventilation: 5 Minutes, 12 Times Daily" (Active Comparator): This arm of the study focuses on a more frequent approach to providing infants with diaper-free air exposure as a method to facilitate healing from diaper dermatitis. In this group, participants experience diaper-free intervals for a duration of 5 minutes, repeated twelve times throughout the day.
  Interventions: Behavioral: Diaper-Free Air Exposure Protocol"

INTERVENTIONS:
Behavioral: Diaper-Free Air Exposure Protocol" — The Diaper-Free Air Exposure Protocol is designed to promote the healing of mild diaper dermatitis in infants through structured periods of diaper-free time. This intervention consists of allowing infants to be without a diaper for specific durations throughout the day, aiming to enhance airflow to the affected area and reduce moisture accumulation, which can exacerbate skin irritation.
  Duration and Frequency: Infants will be exposed to diaper-free intervals lasting 5 minutes each. The intervention will be implemented with varying frequencies based on the study group: 6 times daily for Group A and 12 times daily for Group B.
  Environment: The diaper-free periods will take place in a safe and comfortable environment, ensuring that the infants are not exposed to potential hazards (e.g., cold surfaces, unsanitary conditions). Caregivers will be instructed to monitor the infants during these periods to ensure their safety and comfort.

SUMMARY:
Brief Summary Title: The Effect of Ventilation Frequency on Diaper Dermatitis Recovery and Maternal Self-Efficacy in Infants Aged 0-3 Months: A Randomized Controlled Trial

Authors: Fatma Şule Bilgiç, Aysu Yıldız Karaahmet, Shahla Shafaati Laleh

Background: Diaper dermatitis (DD) is a prevalent condition affecting infants aged 0-3 months, causing discomfort for both infants and parents. While traditional management focuses on skin protection, the role of ventilation in recovery is not well-studied. This trial investigates the impact of different ventilation frequencies on diaper dermatitis healing and maternal self-efficacy.

Methods: A randomized controlled trial included 130 infants with mild diaper dermatitis, divided into two groups: Group A (5 minutes of diaper-free air exposure 6 times a day) and Group B (5 minutes of exposure 12 times a day). Recovery was assessed using the Uncomplicated Diaper Dermatitis Severity Rating Scale (UDDSRSI) and maternal self-efficacy was measured with the Perceived Maternal Self-Efficacy Scale (PMSS).

Keywords: Diaper dermatitis, ventilation, maternal self-efficacy, infant care, randomized controlled trial.

DETAILED DESCRIPTION:
Detailed Description Title: The Effect of Ventilation Frequency on Diaper Dermatitis Recovery and Maternal Self-Efficacy in Infants Aged 0-3 Months: A Randomized Controlled Trial Background: Diaper dermatitis (DD) is a prevalent skin condition in infants, particularly affecting those aged 0-3 months. It is characterized by inflammation, redness, and irritation in the diaper area, which can lead to significant discomfort for the infant and distress for the caregivers. Traditional management strategies focus on skin protection through frequent diaper changes, proper hygiene practices, and the use of barrier creams. However, the potential benefits of increased ventilation in the diaper area have not been sufficiently explored. This study aims to evaluate how varying frequencies of diaper-free air exposure can influence the recovery of diaper dermatitis and the perceived self-efficacy of mothers caring for affected infants.

Methods: A randomized controlled trial was conducted at a private hospital's Pediatric Outpatient Clinic over a year, from January 2023 to January 2024. A total of 130 infants diagnosed with mild diaper dermatitis were recruited and randomly assigned to two intervention groups:

Group A: Received 5 minutes of diaper-free air exposure 6 times a day. Group B: Received 5 minutes of diaper-free air exposure 12 times a day.

Data were collected at baseline and upon resolution of diaper dermatitis using:

Uncomplicated Diaper Dermatitis Severity Rating Scale (UDDSRSI): This scale assesses the severity of diaper dermatitis based on criteria such as erythema, papules, and skin breakdown.

Perceived Maternal Self-Efficacy Scale (PMSS): This scale evaluates mothers' confidence in their caregiving abilities.

Data Collection Process: The study involved a comprehensive data collection process, including a detailed questionnaire about sociodemographic characteristics and infant health status. Mothers were trained on proper diaper cleaning techniques and the importance of ventilation in managing diaper dermatitis through a structured educational session.

Keywords: Diaper dermatitis, ventilation, maternal self-efficacy, infant care, randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged from 0 months (newborn) to 12 months.
* Infants must exhibit mild to moderate diaper dermatitis as assessed by the Modified Diaper Dermatitis Severity Index (MDDSI) at baseline.
* Written informed consent must be obtained from the parent or legal guardian prior to participation in the study.
* Infants must be in overall good health, without any significant medical conditions that would interfere with the study or require additional treatment for skin conditions.

Exclusion Criteria:

* Infants with severe diaper dermatitis or other dermatological conditions affecting the diaper area (e.g., fungal infections, bacterial infections, or other rashes) will be excluded.
* Infants who have received topical treatments (e.g., antifungals, corticosteroids) for diaper dermatitis or other skin conditions within the past 2 weeks prior to enrollment.
* Infants with significant health issues, such as immunosuppression, chronic skin conditions, or other comorbidities that may affect the skin's integrity.
* Infants currently enrolled in other clinical trials or studies that may influence the outcomes of this study.

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Severity of diaper dermatitis in infants measured by the Modified Diaper Dermatitis Severity Index (MDDDSI) | Baseline and weekly assessments for 6 weeks during intervention
  Skin assessments conducted at baseline and weekly using MDDDSI.
  Scoring criteria: erythema, edema, erosion, papules, exudate.
  Each item scored 0-3; higher scores indicate more severe dermatitis.
  Total score used to determine overall severity.

SECONDARY OUTCOMES:
Maternal self-efficacy measured by the Perceived Maternal Self-Efficacy Scale (PMSS) | Maternal self-efficacy will be assessed using the Perceived Maternal Self-Efficacy Scale (PMSS), a validated 20-item 4-point Likert scale (range: 20-80). Higher scores indicate greater perceived maternal self-efficacy. The scale will be administered at b
  Baseline and at dermatitis recovery (average 1-3 days after intervention)

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Zeytinburnu, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No